CLINICAL TRIAL: NCT03490227
Title: Measurement of Body Fat in Infants
Acronym: Baby Fat Pilot
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2017-050
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Brown Adipose Tissue; Body Composition
Keywords: neonates; brown adipose tissue; body composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Up to 10 infants will complete the study aimed to establish a technique for measuring whole body adiposity and brown adipose tissue in infant subjects using dual energy x-ray absorptiometry and magnetic resonance imaging, respectively.

ELIGIBILITY:
Inclusion Criteria:

* healthy, full-term infant
* aged 14-28 days at Visit 1

Exclusion Criteria:

* born preterm (<37 weeks gestation)
* implanted metal or electronic objects that render MRI unsafe
* unable to complete 2 clinic visits 1-10 days apart at Pennington Biomedical Research Center

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Up to 10 healthy, full term infants aged 14 to 28 days old at enrollment with no contraindications to MRI will be recruited to Pennington Biomedical Research Center to participate in this study which includes two study visits to be completed within 1-10 days apart.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This is an observational study where all participants did DXA once and MRI twice in order to assess infant body composition and brown adipose tissue.
Period: Overall Study
Arm/Group | All Participants
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: days] | 22.6 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Gestational Age at Birth [Mean (Standard Deviation); unit: weeks] | 39.129 (1.296)

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Fat Mass
Description: Whole body fat mass will be measured in infant subjects using dual energy x-ray absorptiometry.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of fat mass
Groups:
- All Participants: This is an observational study where all participants did DXA once in order to assess infant body composition.
Arm/Group | All Participants
Number analyzed (Participants) | 10
percentage of fat mass | 20.8 (1.8)

2. Primary Outcome: Average Brown Adipose Tissue Volume at First Visit
Description: Magnetic resonance imaging were traced for lipid: water ratio in the supraclavicular region. Brown adipose tissue volume was calculated by summing all brown adipose tissue volume in the supraclavicular region with a lipid: water ration (or fat signal fraction) between 10-50%.
Time Frame: 1 day
Population: One scan was not analyzed. The scan was completed but did not provide valid data.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Groups:
- All Participants: This is an observational study where all participants did MRI twice in order to assess infant brown adipose tissue volume.
Arm/Group | All Participants
Number analyzed (Participants) | 9
cubic centimeters | 5.41 (0.88)

3. Primary Outcome: Average Brown Adipose Tissue Volume at Second Visit
Description: as for outcome 2
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | All Participants
Number analyzed (Participants) | 10
cubic centimeters | 5.50 (1.30)

4. Secondary Outcome: Average Fat Signal Fraction of Brown Adipose Tissue at First Visit
Description: Magnetic resonance imaging scans were traced for lipid: water ratio in the supraclavicular region. Fat signal fraction is defined as the lipid: water ratio found in the lipid tissues in the supraclavicular region. Only traced lipid tissues (between 10-50%) were included in the average fat signal fraction because only traced lipid tissues were classified as brown adipose tissue.
Time Frame: 1 day
Population: One scan was not analyzed. The scan was completed but did not provide valid data.
Measure: Mean (Standard Deviation); unit: Percentage of lipid
Arm/Group | All Participants
Number analyzed (Participants) | 9
Percentage of lipid | 16.64 (3.31)

5. Secondary Outcome: Average Fat Signal Fraction of Brown Adipose Tissue at Second Visit
Description: as for outcome 4
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Percentage of lipid
Arm/Group | All Participants
Number analyzed (Participants) | 10
Percentage of lipid | 16.43 (3.41)

6. Secondary Outcome: Reliability of Average Brown Adipose Tissue Volume Measurement Between the First and Second Visit
Description: Reliability of average brown adipose tissue volume measurement between visits was determined using intraclass correlation coefficient. Paired average brown adipose tissue volume measurements were included in the intraclass correlation coefficient computation.
Time Frame: 2 days within 10 days apart
Population: One scan was not analyzed. The scan was completed but did not provide valid data.
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient
Groups:
- All Participants: This is an observational study where all participants did MRI twice in order to assess the reliability of measuring brown adipose tissue in infants.
Arm/Group | All Participants
Number analyzed (Participants) | 9
intraclass correlation coefficient | 0.92 [0.65 to 0.98]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=10)
Flatulence (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
During one MRI scan occurring at the respective participant's first visit, a magnetic resonance imaging (MRI) machine malfunction led to acquisition of images that were unanalyzable and therefore unusable.

The study is limited by a small and relatively homogenous sample of ten infants. Given the nature of the method development study, we did not enroll equal numbers of males and females.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03490227/Prot_SAP_000.pdf